CLINICAL TRIAL: NCT03875092
Title: A Randomized, Double-Blind, Phase III Study of Carboplatin-Paclitaxel/Nab-Paclitaxel Chemotherapy With or Without Pembrolizumab (MK-3475) in First Line Metastatic Squamous Non-small Cell Lung Cancer Subjects (KEYNOTE-407)
Brief Title: A Study of Carboplatin-Paclitaxel/Nab-Paclitaxel Chemotherapy With or Without Pembrolizumab (MK-3475) in Adults With First Line Metastatic Squamous Non-small Cell Lung Cancer (MK-3475-407/KEYNOTE-407)-China Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-407 China Extension; 173568 (Registry Identifier: JAPIC-CTI); MK-3475-407 (Other: MSD Protocol Number); KEYNOTE-407 (Other: MSD)
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Results first posted 2021-10-20 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Chemotherapy (Experimental): Participants receive pembrolizumab 200 mg by intravenous (IV) infusion prior to chemotherapy on Day 1 of each 21-day cycle for up to 35 cycles PLUS paclitaxel (200 mg/m^2 by IV infusion on Day 1 of each 21-day cycle for 4 cycles) PLUS carboplatin Area Under the Curve (AUC) 6 by IV infusion on Day 1 of each 21-day cycle for 4 cycles.
  Interventions: Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin
- Chemotherapy (Active Comparator): Participants receive normal saline by IV infusion prior to chemotherapy on Day 1 of each 21-day cycle for up to 35 cycles PLUS paclitaxel (200 mg/m^2 by IV infusion on Day 1 of each 21-day cycle for 4 cycles) PLUS carboplatin AUC 6 by IV infusion on Day 1 of each 21-day cycle for 4 cycles.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Saline placebo for pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab + Chemotherapy
Drug: Paclitaxel — IV infusion
  Other Names: TAXOL®
Drug: Carboplatin — IV infusion Carboplatin dose should not exceed 900 mg.
  Other Names: PARAPLATIN®
Drug: Saline placebo for pembrolizumab — IV infusion
  Arms: Chemotherapy

SUMMARY:
In this China extension study, carboplatin and paclitaxel with or without pembrolizumab (MK-3475, KEYTRUDA®) will be administered to Chinese adults with first line metastatic squamous non-small cell lung cancer (NSCLC).

The primary hypotheses are that treatment with pembrolizumab prolongs: 1) Progression-free Survival (PFS) by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by a blinded central imaging vendor compared to placebo, and 2) Overall Survival (OS) in Chinese participants.

After analysis of interim results was conducted, the protocol was amended (Amendment 5) to allow participants the option to discontinue placebo in the control arm and to switch to pembrolizumab in the event of documented progressive disease as assessed by central review.

DETAILED DESCRIPTION:
The MK-3475-407-China Extension Study enrolled a total of 125 participants, of which 15 participants have been also previously enrolled in the MK-3475-407 global study (NCT02775435). This China extension study did not include nano particle albumin-bound paclitaxel (nab-paclitaxel) that was an option in the global base study, because nab-paclitaxel it is not yet approved for treatment of NSCLC in China.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of stage IV (M1a or M1b-American Joint Committee on Cancer [AJCC]) squamous NSCLC.
* Has measurable disease based on RECIST 1.1 as determined by the local site investigator/radiology assessment.
* Has not received prior systemic treatment for metastatic NSCLC.
* Has provided tumor tissue from locations not radiated prior to biopsy.
* Has a life expectancy of at least 3 months.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* Has adequate organ function.
* If female of childbearing potential, is willing to use an adequate method of contraception for the course of the study through 180 days after the last dose of study treatment.
* If male with a female partner(s) of child-bearing potential, must agree to use an adequate method of contraception starting with the first dose of study treatment through 95 days after the last dose of study treatment. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

Exclusion Criteria:

* Has non-squamous histology NSCLC.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to administration of pembrolizumab.
* Before the first dose of study drug: a) Has received prior systemic cytotoxic chemotherapy for metastatic disease; b) Has received other targeted or biological antineoplastic therapy (e.g., erlotinib, crizotinib, cetuximab) for metastatic disease; c) Has had major surgery (<3 weeks prior to first dose).
* Received radiation therapy to the lung that is >30 Gray (Gy) within 6 months of the first dose of study treatment.
* Completed palliative radiotherapy within 7 days of the first dose of study treatment.
* Is expected to require any other form of antineoplastic therapy while on study.
* Has received a live-virus vaccination within 30 days of planned treatment start.
* Has a known history of prior malignancy except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has pre-existing peripheral neuropathy that is ≥ Grade 2 by Common Terminology Criteria for Adverse Events (CTCAE) Version 4 criteria.
* Previously had a severe hypersensitivity reaction to treatment with another monoclonal antibody.
* Has a known sensitivity to any component of carboplatin or paclitaxel or nab-paclitaxel.
* Has active autoimmune disease that has required systemic treatment in past 2 years.
* Is on chronic systemic steroids.
* Had prior treatment with any other anti-programmed cell death 1 (anti-PD-1), or programmed cell death ligand 1 (PD-L1) or PD-L2 agent or an antibody or a small molecule targeting other immuno-regulatory receptors or mechanisms.
* Has participated in any other pembrolizumab trial and has been treated with pembrolizumab.
* Has an active infection requiring therapy.
* Has known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection.
* Is, at the time of providing documented informed consent, a regular user (including "recreational use") of any illicit drugs or has a recent history (within the last year) of substance abuse (including alcohol).
* Has interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Cheng Y, Zhang L, Hu J, Wang D, Hu C, Zhou J, Wu L, Cao L, Liu J, Zhang H, Sun H, Wang Z, Gao H, Sun Y, Li B, Hu X, Schwarzenberger P, Paz-Ares L. Pembrolizumab Plus Chemotherapy for Chinese Patients With Metastatic Squamous NSCLC in KEYNOTE-407. JTO Clin Res Rep. 2021 Sep 25;2(10):100225. doi: 10.1016/j.jtocrr.2021.100225. eCollection 2021 Oct. PMID 34661177
- [Derived] Cheng Y, Yang JC, Okamoto I, Zhang L, Hu J, Wang D, Hu C, Zhou J, Wu L, Cao L, Liu J, Zhang H, Sun H, Wang Z, Gao H, Yan Y, Xiao S, Lin J, Pietanza MC, Kurata T. Pembrolizumab plus chemotherapy for advanced non-small-cell lung cancer without tumor PD-L1 expression in Asia. Immunotherapy. 2023 Sep;15(13):1029-1044. doi: 10.2217/imt-2023-0043. Epub 2023 Jul 19. PMID 37465924
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The China extension study included participants previously enrolled in China in the global study for MK-3475-407 (NCT02775435) plus those enrolled during the China extension enrollment period.
Groups:
- Pembrolizumab + Chemotherapy: Participants received pembrolizumab 200 mg by intravenous (IV) infusion prior to chemotherapy on Day 1 of each 21-day cycle for up to 35 cycles PLUS paclitaxel (200 mg/m^2 by IV infusion on Day 1 of each 21-day cycle for 4 cycles) PLUS carboplatin Area Under the Curve (AUC) 6 by IV infusion on Day 1 of each 21-day cycle for 4 cycles.
- Chemotherapy: Participants received normal saline by IV infusion prior to chemotherapy on Day 1 of each 21-day cycle for up to 35 cycles PLUS paclitaxel (200 mg/m^2 by IV infusion on Day 1 of each 21-day cycle for 4 cycles) PLUS carboplatin AUC 6 by IV infusion on Day 1 of each 21-day cycle for 4 cycles.
Period: Overall Study
Arm/Group | Pembrolizumab + Chemotherapy | Chemotherapy
Started | 65 | 60
Treated | 65 | 60
Switched to Pembrolizumab+Chemotherapy | 0 | 38
Received Second Course of Pembrolizumab | 6 | 0
Completed | 0 | 0
Not Completed | 65 | 60
Not completed — Adverse Event | 2 | 5
Not completed — Death | 44 | 51
Not completed — Participation Was Terminated By Sponsor | 19 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Chemotherapy | Chemotherapy | Total
Number analyzed (Participants) | 65 | 60 | 125
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (8.7) | 61.5 (9.1) | 61.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 62 | 57 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 65 | 60 | 125
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 65 | 60 | 125
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Programmed Cell Death-Ligand 1 (PD-L1) Tumor Expression Level: Tumor Proportion Score (TPS) [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. Participants with a TPS ≥1% were classified as PD-L1 positive and participants with a TPS <1% were classified as not PD-L1 positive.
  Participants
    TPS <1% | 25 | 23 | 48
    TPS ≥1% | 37 | 35 | 72
    Unknown | 3 | 2 | 5
Taxane Chemotherapy [Count of Participants; unit: Participants] — Participants were classified according to their taxane chemotherapy regimen: paclitaxel or nab-paclitaxel.
  Participants
    +Paclitaxel | 65 | 60 | 125
    +Nab-paclitaxel | 0 | 0 | 0
Geographic Region [Count of Participants; unit: Participants] — Participants were classified according to their geographic region: East Asia vs. non-East Asia.
  Participants
    East Asia | 65 | 60 | 125
    Non-East Asia | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per Response Criteria in Solid Tumors version 1.1 (RECIST 1.1), PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Note: The appearance of ≥1 new lesions was also considered PD. PFS as assessed by blinded independent central review per RECIST 1.1 is presented. Data are from the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 33 months
Population: The Intent-To-Treat population consisted of all randomized participants, regardless of whether or not they received study treatment. Participants were included in the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy | Chemotherapy
Number analyzed (Participants) | 65 | 60
Months | 8.3 [6.2 to 10.5] | 4.2 [4.0 to 5.4]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy vs Chemotherapy; Test type: Other; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.24 to 0.52] — Based on unstratified Cox regression model with treatment as a covariate, due to small sample size

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. OS is presented. Data are from the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 39 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy | Chemotherapy
Number analyzed (Participants) | 65 | 60
Months | 30.1 [18.2 to NA] — NA=OS upper limit not reached | 12.7 [9.4 to 17.3]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy vs Chemotherapy; Test type: Other; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.28 to 0.70] — Based on unstratified Cox regression model with treatment as a covariate, due to small sample size

3. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed by RECIST 1.1. ORR as assessed by blinded independent central review per RECIST 1.1 is presented.
Time Frame: Up to approximately 33 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Chemotherapy | Chemotherapy
Number analyzed (Participants) | 65 | 60
Percentage of Participants | 80.0 [68.2 to 88.9] | 43.3 [30.6 to 56.8]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy vs Chemotherapy; Test type: Other; Difference in Percentage = 36.7, 95% CI 2-sided [19.9 to 51.6] — Based on unstratified Miettinen & Nurminen method, due to small sample size

4. Secondary Outcome: Duration of Response (DOR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: For participants who demonstrated a confirmed response (Complete Response [CR]: Disappearance of all target lesions or Partial Response [PR]: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until disease progression as assessed by RECIST 1.1 or death. DOR as assessed by blinded independent central review per RECIST 1.1 is presented.
Time Frame: Up to approximately 30 months
Population: The Intent-To-Treat population consisted of all randomized participants, regardless of whether or not they received study treatment, who demonstrated a confirmed response (CR or PR). Participants were included in the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy | Chemotherapy
Number analyzed (Participants) | 65 | 60
Months | 7.1 [4.9 to 14.4] | 3.5 [2.8 to 4.9]

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment. The number of participants who experienced an AE is presented. Data are from the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 31 months
Population: The Safety population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Chemotherapy | Chemotherapy
Number analyzed (Participants) | 65 | 60
Participants | 65 | 60

6. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 29 months
Population: The Safety population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Chemotherapy | Chemotherapy
Number analyzed (Participants) | 65 | 60
Participants | 8 | 4

ADVERSE EVENTS:
Time Frame: All-Cause mortality: Up to 1948 days Adverse events: Up to 1625 days
Description: Mortality data were collected for all randomized participants. Adverse event (AE) data were collected for all participants who received ≥1 dose of study treatment. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Therefore Medical Dictionary for Regulatory Activities (MedDRA) terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment are excluded as AEs.
Groups:
- Chemotherapy > Pembrolizumab Switch Over: Eligible participants with documented disease progression following chemotherapy in "Chemotherapy" arm switched over to receive pembrolizumab 200 mg IV Q3W for up to 35 administrations (approximately 2 years).
- Pembrolizumab > Pembrolizumab Second Course: Eligible participants who received pembrolizumab as a first course (200 mg IV Q3W for up to 35 administrations) and stopped the first course of pembrolizumab due to complete response; or completed the first course of pembrolizumab and had stable disease, partial response, or complete response; but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (approximately 1 year additional).
Arm/Group | Pembrolizumab + Chemotherapy | Chemotherapy | Chemotherapy > Pembrolizumab Switch Over | Pembrolizumab > Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 41/65 | 22/60 | 34/38 | 5/6
Serious Adverse Events (participants affected / at risk) | 35/65 | 22/60 | 10/38 | 0/6
Other Adverse Events (participants affected / at risk) | 65/65 | 60/60 | 32/38 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Chemotherapy (N=65) | Chemotherapy (N=60) | Chemotherapy > Pembrolizumab Switch Over (N=38) | Pembrolizumab > Pembrolizumab Second Course (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 3 (3) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (8) | 5 (5) | 5 (6) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Chemotherapy (N=65) | Chemotherapy (N=60) | Chemotherapy > Pembrolizumab Switch Over (N=38) | Pembrolizumab > Pembrolizumab Second Course (N=6)
Anaemia (Blood and lymphatic system disorders) | 42 (103) | 46 (85) | 11 (17) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 12 (49) | 7 (32) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (6) | 3 (4) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 12 (16) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 8 (15) | 1 (1) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 16 (20) | 14 (21) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 11 (23) | 6 (11) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 24 (42) | 13 (22) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 15 (26) | 10 (12) | 2 (2) | 0 (0)
Asthenia (General disorders) | 10 (16) | 7 (9) | 3 (3) | 0 (0)
Chest discomfort (General disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 4 (4) | 9 (10) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (13) | 3 (8) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 8 (9) | 8 (9) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 12 (14) | 9 (10) | 3 (4) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (6) | 3 (4) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 7 (8) | 6 (7) | 4 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (12) | 3 (5) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 24 (40) | 17 (26) | 6 (7) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 19 (33) | 13 (21) | 3 (3) | 1 (1)
Bilirubin conjugated increased (Investigations) | 3 (18) | 4 (5) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 4 (9) | 2 (3) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 7 (15) | 3 (4) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 5 (26) | 4 (5) | 3 (5) | 1 (2)
Blood chloride decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood cholinesterase decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 4 (11) | 4 (4) | 3 (5) | 2 (5)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 2 (4) | 1 (1) | 2 (3) | 1 (1)
Blood uric acid increased (Investigations) | 5 (16) | 3 (3) | 1 (2) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 10 (12) | 11 (14) | 5 (7) | 1 (2)
Neutrophil count decreased (Investigations) | 50 (195) | 43 (128) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1) | 5 (6) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 16 (53) | 22 (37) | 1 (3) | 1 (2)
Prealbumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 9 (9) | 11 (13) | 3 (3) | 1 (1)
Weight increased (Investigations) | 8 (11) | 2 (2) | 2 (4) | 0 (0)
White blood cell count decreased (Investigations) | 51 (192) | 42 (131) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 4 (5) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 25 (43) | 19 (25) | 5 (5) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (20) | 7 (13) | 6 (9) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 10 (31) | 3 (5) | 6 (7) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (12) | 13 (18) | 5 (5) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (9) | 1 (1) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 6 (8) | 4 (5) | 2 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 16 (34) | 12 (20) | 6 (8) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (8) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (18) | 10 (14) | 6 (7) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (43) | 14 (19) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (8) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (19) | 8 (10) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (17) | 13 (13) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 29 (46) | 22 (25) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 6 (6) | 8 (8) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 6 (7) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 10 (14) | 2 (3) | 3 (4) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4) | 4 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 7 (10) | 4 (5) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 12 (16) | 3 (6) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 11 (18) | 3 (6) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 3 (3) | 0 (0)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 51 (53) | 40 (40) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 16 (25) | 3 (4) | 3 (4) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 2 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (2):
  • Study Protocol (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT03875092/Prot_002.pdf
  • Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT03875092/SAP_003.pdf